CLINICAL TRIAL: NCT00004264
Title: Phase I/II Trial of Amifostine, High-Dose Cisplatin and Docetaxel in Patients With Advanced Lung Cancer
Brief Title: Docetaxel, Cisplatin, and Amifostine in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067523; WCCC-CO-9653; NCI-G00-1668
Record Dates: First submitted 2000-01-28; First posted 2004-07-26 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-08

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Amifostine; Cisplatin; Docetaxel

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of combining docetaxel, cisplatin, and amifostine in treating patients who have advanced non-small cell lung cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of docetaxel when combined with amifostine and high dose cisplatin in patients with advanced non-small cell lung cancer. II. Determine the response rate and survival of these patients treated with this regimen. III. Determine the tolerability of this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study of docetaxel. Patients receive amifostine IV over 15 minutes, immediately followed by docetaxel IV over 1 hour, followed at hour 2 by amifostine as above, immediately followed by high dose cisplatin IV over 30 minutes. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of patients receive escalating doses of docetaxel until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unresectable advanced non-small cell lung cancer Stable CNS metastases allowed

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: AST no greater than 2.5 times upper limit of normal (ULN) AND alkaline phosphatase no greater than ULN OR AST no greater than ULN AND alkaline phosphatase no greater than 4 times ULN Renal: Creatinine clearance at least 60 mL/min Other: Not pregnant Fertile patients must use effective contraception No peripheral neuropathy worse than grade 1

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Any type and any number of prior chemotherapy regimens allowed and recovered Greater than 3 months since prior cisplatin and recovered Endocrine therapy: Prior endocrine therapy allowed and recovered Radiotherapy: Prior radiotherapy allowed and recovered Surgery: Prior surgery allowed and recovered Other: No other concurrent medications which could cause renal injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States